CLINICAL TRIAL: NCT01158391
Title: Trial of Patterned Oral Somatosensory Entrainment
Brief Title: Trial of Patterned Oral Somatosensory Entrainment for Shortening Time to Oral Feeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KC BioMediX, Inc (Industry)
Collaborators: Innara Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC_BMDX_002
Record Dates: First submitted 2010-06-24; First posted 2010-07-08 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Infant, Extremely Premature; Length of Stay; Feeding
Keywords: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NTrainer® Intervention (Experimental): NTrainer® Intervention - Infants in the experimental group will receive the NTrainer System patterned synthetic orocutaneous stimulation during the first 30 minutes of a tube (gavage) feeding session. The intervention may be provided up to 4 times daily to achieve an average of 30 sessions distributed over a two week period.
  Interventions: Device: NTrainer® Intervention
- Control Intervention (Sham Comparator): Control Intervention - Infants in the Control group will be provided orocutaneous stimulation with a 'quiet pacifier' during the first 30 minutes of a tube (gavage) feeding session. The intervention may be provided up to 4 times daily to achieve an average of 30 sessions distributed over a two week period.
  Interventions: Device: Control Intervention

INTERVENTIONS:
Device: NTrainer® Intervention
  Other Names: KC BioMedix NTrainer; NTrainer System; Actifier
  Arms: NTrainer® Intervention
Device: Control Intervention
  Other Names: Non-nutritive Sucking; NNS Opportunity
  Arms: Control Intervention

SUMMARY:
The primary hypothesis is that the preterm infants (26 0/7 to 30 6/7 weeks gestational age) who undergo the NTrainer System® training will transition to full oral feeds faster than the control group (i.e. the study group will be superior to the control).

The secondary hypothesis is that the infants in the NTrainer System® experimental group will have shorter lengths of stay.

DETAILED DESCRIPTION:
Patterned Oral Somatosensory Intervention

The interventions (Treatment vs Control) will be initiated simultaneously with tube (gavage) feeds as early as 30 weeks post-menstrual age. Before and during each training session the infant will be evaluated for the following criteria:

Criteria for Initiation of each intervention:

1. Not on continuous vasopressor medications
2. Feeding in previous 48 hours.
3. Not mechanically ventilated. If the infant is on CPAP or Nasal cannula >2 liters per minute, then the FiO2 must be <40%.

Criteria for Exiting an Intervention Session:

1. If during an intervention the baby experiences Apnea/Bradycardic/Desaturation events requiring nursing stimulation or intervention during the training--hold future interventions for one session.
2. If the interventions are held for 3 consecutive sessions, hold interventions for a full day (24 hours).
3. If interventions are held for 3 days (72 hours) and if GA is <32 weeks when ready to restart therapy sessions, then complete another 10 days of interventions.
4. If interventions are held for 3 days (72 hours) and if GA is >32 weeks when ready to restart therapy, then complete the remaining N interventions sessions for a total of 10 days of therapy.
5. If interventions are held for 3 days (72 hours) and the infant is on full oral feeds when ready to restart therapy interventions then discontinue any remaining interventions sessions.

The Interventions

Infants in the Treatment and Control group will receive orocutaneous stimulation up to four times daily during the first 30 minutes of a tube (gavage) feeding session to achieve an average of 30 therapy sessions distributed over a two week period.

Infants assigned to the either group will be offered the pacifier by gently placing the pacifier on the lips. The pacifier should not be forced into the mouth and should not be moved in any manner that would represent any form of patterned input such as moving the pacifier in and out, tapping on the lips or face or massaging the mouth or oral facial structure.

All other preparatory, infant positioning, and sampling conditions will be equal among groups. The healthcare team will continue to promote feeding and growth at the standard of care for babies in both groups.

Treatment Group

Infants in the Treatment group will receive the NTrainer System® patterned synthetic orocutaneous stimulation. A single NTrainer intervention runs for 20 minutes and involves three 3 minute sessions during which the pacifier pulses. The pulsing sessions are separated by 5.5 min breaks where the pacifier is quiet.

Control Group

Infants assigned to the control group will receive an orocutaneous intervention in which the infant will be offered a 20 minute non-nutritive sucking opportunity with a 'quiet' pacifier.

Breast Feeding Non-nutritive breastfeeding and nutritive breastfeeding practice will not be altered or changed by the interventions. The availability of the mother will be taken into consideration for the scheduling of any intervention sessions and no study intervention will interfere with breastfeeding behavior.

Safety To help ensure the safety of the study participants the heart rate, oxygen saturation, and blood pressure will be monitored throughout the therapy session.

ELIGIBILITY:
Inclusion Criteria

- Birth Gestational age 26 0/6 - 30 6/7 weeks

Exclusion Criteria

* Chromosomal abnormalities
* Congenital anomalies included but not limited to
* craniofacial malformation
* cyanotic congenital heart disease
* gastroschisis
* omphalocele
* diaphragmatic hernia or other major gastrointestinal anomalies
* Major neurological anomaly
* Infants with history of surgical necrotizing enterocolitis (stage III)
* Infants with vocal cord paralysis
* Infants with neonatal seizures
* Infants with meningitis at time of enrollment
* Infants who are nippling all feeds at the time of enrollment
* Infants with narcotic abstinence syndrome (NAS)
* Infants enrolled in another clinical study

Ages: 26 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2010-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The length of time to reach 100% full oral feeds | 14 days on average
  Time (in days) from initiation of oral feedings to the first oral intake that results in 100% oral feeding (definition of 100% oral feeding: no gavage supplementation and taking at least 120 milliliters per kilogram per day for 48 consecutive hours of breast milk, fortified breast milk or preterm formula as ordered by the child's physician.

SECONDARY OUTCOMES:
The reduction in length of stay as a result of therapy | 24 days on average
  The difference in length of hospital stay (days) between experimental and control.

CONTACTS AND LOCATIONS:
Overall Officials: Dongli Song, MD, Principal Investigator — Santa Clara Valley Medical Center
Locations (5):
- United States (5):
  - Santa Clara Valleye Medical Center, San Jose, California
  - Montefiore Medical Center Weiler Hopsital, The Bronx, New York
  - Montefiore Medical Center - Wakefield Hopsital, The Bronx, New York
  - Cook Children's Medical Center, Fort Worth, Texas
  - North Central Baptist Hospital, San Antonio, Texas

REFERENCES:
- [Derived] Song D, Jegatheesan P, Nafday S, Ahmad KA, Nedrelow J, Wearden M, Nemerofsky S, Pooley S, Thompson D, Vail D, Cornejo T, Cohen Z, Govindaswami B. Patterned frequency-modulated oral stimulation in preterm infants: A multicenter randomized controlled trial. PLoS One. 2019 Feb 28;14(2):e0212675. doi: 10.1371/journal.pone.0212675. eCollection 2019. PMID 30817764